CLINICAL TRIAL: NCT00309985
Title: CHAARTED: ChemoHormonal Therapy Versus Androgen Ablation Randomized Trial for Extensive Disease in Prostate Cancer
Brief Title: Androgen Ablation Therapy With or Without Chemotherapy in Treating Patients With Metastatic Prostate Cancer
Acronym: CHAARTED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3805; E3805 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
Keywords: metastatic hormone-sensitive prostate cancer; docetaxel
MeSH Terms: interventions — Androgen Antagonists; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Androgen-Deprivation Therapy and Docetaxel (Experimental): Patients receive androgen-deprivation therapy (including luteinizing hormone-releasing hormone [LHRH] agonist therapy, LHRH antagonist therapy, or surgical castration). Patients also receive docetaxel IV over 1 hour on day 1. Treatment with docetaxel repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: androgen-deprivation therapy; Drug: docetaxel
- Androgen-Deprivation Therapy alone (Active Comparator): Patients receive androgen-deprivation therapy (including luteinizing hormone-releasing hormone [LHRH] agonist therapy, LHRH antagonist therapy, or surgical castration) alone.
  Interventions: Drug: androgen-deprivation therapy

INTERVENTIONS:
Drug: androgen-deprivation therapy — LHRH analogs are administered with a variety of techniques such as subcutaneously, intramuscularly, or insertion, while antiandrogens (flutamide and bicalutamide) were given orally.
Drug: docetaxel — Given IV
  Other Names: Taxotere; RP 56976; NSC #628503
  Arms: Androgen-Deprivation Therapy and Docetaxel

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Androgen ablation therapy may stop the adrenal glands from making androgens. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether androgen-ablation therapy is more effective with or without docetaxel in treating metastatic prostate cancer.

PURPOSE: This randomized phase III trial is studying androgen-ablation therapy and chemotherapy to see how well they work compared to androgen-ablation therapy alone in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the ability of early chemotherapy to improve overall survival of patients commencing androgen deprivation for metastatic prostate cancer.

Secondary

* Determine whether early chemotherapy can increase the time to clinical progression (radiographic or symptomatic deterioration due to disease) over hormonal therapy alone.
* Determine whether early chemotherapy can increase the time to development of hormone-refractory disease over hormonal therapy alone.
* Determine whether early chemotherapy can increase the time to serological progression over hormonal therapy alone.
* Determine rates of biochemical response at 6 months and 12 months in the chemohormonal arm versus the hormonal therapy alone arm.
* Determine the frequency of adverse events and the tolerability of chemotherapy combined with hormonal therapy versus hormonal therapy alone.
* Determine whether the postulated clinically meaningful increase in disease control is associated with an alteration in overall quality of life using the Functional Assessment of Cancer Therapy-Prostate questionnaire.
* Determine the ability of prostate-specific antigen (PSA) changes to be a surrogate for clinical benefit from therapy and overall survival.

Tertiary

* Determine whether there are proteins differentially translated from the genome in hormone-sensitive prostate cancer, prostate cancer that has responded to hormonal therapy, and hormone-refractory prostate cancer.
* Determine the frequency of constitutive polymorphisms of enzymes involved in steroid metabolism and other carcinogenic processes.
* Determine whether the amount and frequency of certain carcinogenic proteins in prostate cancer tissue such as C-X-C chemokine receptor type 4 (CXCR-4) and manganese superoxide dismutase can be correlated with a poor prognosis.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (≥ 70 vs < 70), ECOG performance status (0-1 vs 2), combined androgen blockade for > 30 days (yes vs no), duration of prior adjuvant hormonal therapy (> 12 months vs ≤ 12 months), concurrent bisphosphonate use (yes vs no), and volume of disease (low vs high). Patients are randomized to 1 of 2 treatment arms.

* Arm A (Androgen-Deprivation Therapy and Docetaxel): Patients receive androgen-deprivation therapy (including luteinizing hormone-releasing hormone [LHRH] agonist therapy, LHRH antagonist therapy, or surgical castration). Patients also receive docetaxel intravenously (IV) over 1 hour on day 1. Treatment with docetaxel repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm B (Androgen-Deprivation Therapy alone): Patients receive androgen-deprivation therapy (as in arm A) alone.

Quality of life is assessed at baseline and at months 3, 6, 9 and 12.

After completion of study treatment, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer
* Metastatic disease
* On androgen-deprivation therapy for < 120 days
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2

  * PS 2 eligible only if decline in PS is due to metastatic prostate cancer
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ upper limit of normal (ULN)
* Alanine aminotransferase (ALT) ≤ 2.5 times ULN
* Creatinine clearance ≥ 30 mL/min
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 times ULN (unless on therapeutic anticoagulation)
* Partial thromboplastin time (PTT) ≤ 1.5 times ULN (unless on therapeutic anticoagulation)
* Fertile patients must use effective contraception
* At least 4 weeks since prior major surgery and recovered from all toxicity prior to randomization
* Prior adjuvant or neoadjuvant hormonal therapy allowed provided the following are true:

  * Therapy was discontinued ≥ 12 months ago AND there is no evidence of disease, as defined by 1 of the following:

    * PSA < 0.1 ng/dL after prostatectomy plus hormonal therapy
    * PSA < 0.5 ng/dL and has not doubled above nadir after radiotherapy plus hormonal therapy
  * Therapy lasted no more than 24 months

    * Last depot injection must have expired by the 24-month mark
* Prior palliative radiotherapy allowed if commenced within 30 days before starting androgen deprivation
* Anti-androgen therapy allowed as single-agent therapy ≤ 7 days before medial castration to prevent flare
* More than 30 days (or 6 half-lives) (whichever is longer) since prior participation in another clinical trial
* Concurrent participation in nontherapeutic trials allowed
* Concurrent antiandrogen therapy (e.g., bicalutamide or flutamide) allowed, but not as sole hormonal therapy

Exclusion Criteria:

* Prostate-specific antigen (PSA) level has risen and met criteria for progression from its lowest point between the start of androgen-deprivation therapy and randomization
* Prior malignancy in the past 5 years except for basal cell or squamous cell carcinoma of the skin

  * Other malignancies that are considered to have low potential to progress (e.g., grade 2, T1a transitional cell carcinoma) may be allowed if approved by study chair
* Peripheral neuropathy > grade 1
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Active cardiac disease, including the following:

  * Active angina
  * Symptomatic congestive heart failure
  * Myocardial infarction within the past 6 months
* Prior chemotherapy in adjuvant or neoadjuvant setting
* Prior hormone therapy in the metastatic setting
* Concurrent 5-alpha reductase inhibitors
* Simultaneous enrollment on Cancer and Leukemia Group B (CALGB) 90202

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2006-09-26 (Actual); Primary Completion 2013-12-23 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, MBBS, Study Chair — Dana-Farber Cancer Institute
Locations (343):
- United States (343):
  - Providence Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Mather Veteran Affairs Medical Center, Mather, California
  - Mercy Cancer Center at Mercy Medical Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Saint Helena Hospital, St. Helena, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center, Vallejo, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute at St. Luke's, Twin Falls, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Cottage, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology-Oncology Associates at Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Quincy, Quincy, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer. N Engl J Med. 2015 Aug 20;373(8):737-46. doi: 10.1056/NEJMoa1503747. Epub 2015 Aug 5. PMID 26244877
- [Derived] Guo S, Zhang J, Halabi S. Joint Modelling of Longitudinal Measurements and Time-to-Event Outcomes With a Cure Fraction Using Functional Principal Component Analysis. Stat Med. 2024 Dec 30;43(30):6059-6072. doi: 10.1002/sim.10289. Epub 2024 Dec 5. PMID 39633601
- [Derived] Lage DE, Michaelson MD, Lee RJ, Greer JA, Temel JS, Sweeney CJ. Outcomes of older men receiving docetaxel for metastatic hormone-sensitive prostate cancer. Prostate Cancer Prostatic Dis. 2021 Dec;24(4):1181-1188. doi: 10.1038/s41391-021-00389-2. Epub 2021 May 18. PMID 34007017
- [Derived] Martini A, Pfail J, Montorsi F, Galsky MD, Oh WK. Surrogate endpoints for overall survival for patients with metastatic hormone-sensitive prostate cancer in the CHAARTED trial. Prostate Cancer Prostatic Dis. 2020 Dec;23(4):638-645. doi: 10.1038/s41391-020-0231-5. Epub 2020 Apr 20. PMID 32313142
- [Derived] Morgans AK, Chen YH, Sweeney CJ, Jarrard DF, Plimack ER, Gartrell BA, Carducci MA, Hussain M, Garcia JA, Cella D, DiPaola RS, Patrick-Miller LJ. Quality of Life During Treatment With Chemohormonal Therapy: Analysis of E3805 Chemohormonal Androgen Ablation Randomized Trial in Prostate Cancer. J Clin Oncol. 2018 Apr 10;36(11):1088-1095. doi: 10.1200/JCO.2017.75.3335. Epub 2018 Mar 9. PMID 29522362
- [Derived] Kyriakopoulos CE, Chen YH, Carducci MA, Liu G, Jarrard DF, Hahn NM, Shevrin DH, Dreicer R, Hussain M, Eisenberger M, Kohli M, Plimack ER, Vogelzang NJ, Picus J, Cooney MM, Garcia JA, DiPaola RS, Sweeney CJ. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer: Long-Term Survival Analysis of the Randomized Phase III E3805 CHAARTED Trial. J Clin Oncol. 2018 Apr 10;36(11):1080-1087. doi: 10.1200/JCO.2017.75.3657. Epub 2018 Jan 31. PMID 29384722
- [Derived] Harshman LC, Chen YH, Liu G, Carducci MA, Jarrard D, Dreicer R, Hahn N, Garcia JA, Hussain M, Shevrin D, Eisenberger M, Kohli M, Plimack ER, Cooney M, Vogelzang NJ, Picus J, Dipaola R, Sweeney CJ; ECOG-ACRIN 3805 Investigators. Seven-Month Prostate-Specific Antigen Is Prognostic in Metastatic Hormone-Sensitive Prostate Cancer Treated With Androgen Deprivation With or Without Docetaxel. J Clin Oncol. 2018 Feb 1;36(4):376-382. doi: 10.1200/JCO.2017.75.3921. Epub 2017 Dec 20. PMID 29261442
- [Derived] Scott E. Chemohormonal therapy in metastatic hormone-sensitive prostate cancer. Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Department of Medicine; Department of Biostatistics and Computational Biology; Dana-Farber Cancer Institute, Boston; Harvard Medical School, Boston; Johns Hopkins University, Baltimore; University of Wisconsin Carbone Cancer Center; School of Medicine and Public Health; Madison; Fox Chase Cancer Center, Temple University Health System, Philadelphia; Indiana University Melvin and Bren Simon Cancer Center, Indianapolis; Mayo Clinic, Rochester, MN; University Hospitals Case Medical Center, Seidman Cancer Center; Cleveland Clinic Taussig Cancer Institute; Both in Cleveland; University of Virginia Cancer Center, Charlottesville; Comprehensive Cancer Centers of Nevada, Las Vegas; Siteman Cancer Center, Washington University School of Medicine, St. Louis; NorthShore University Health System, Evanston, IL; University of Michigan Comprehensive Cancer Center, Ann Arbor; Rutgers Cancer Institute of New Jersey, New Brunswick.N Engl J Med. 2015 Aug 20;373(8):737-46. [Epub 2015 Aug 5]. doi: 10.1056/NEJMoa1503747. Urol Oncol. 2017 Mar;35(3):123. doi: 10.1016/j.urolonc.2016.12.021. Epub 2017 Feb 1. PMID 28159490
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on July 28, 2006, accrued its first patient on September 26, 2006, and closed to accrual on November 21, 2012, after accrual of 790 patients.
Groups:
- Androgen-Deprivation Therapy Alone: Patients receive androgen-deprivation therapy (including luteinizing hormone-releasing hormone [LHRH] agonist therapy, LHRH antagonist therapy, or surgical castration).
Period: Overall Study
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Started | 397 | 393
Toxicity Analysis | 390 | 392
Both Baseline and 3-month FACT-P Evals | 334 | 299
Completed | 335 | 392 (Arm B tx info was not collected so only 1 patient w/o follow-up data was considered "not completed".)
Not Completed | 62 | 1
Not completed — Disease progression | 12 | 0
Not completed — Adverse Event | 30 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Never started treatment | 7 | 0
Not completed — Complicating disease | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Chemotherapy discontinued only | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone | Total
Number analyzed (Participants) | 397 | 393 | 790
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 88] | 63 [39 to 91] | 63 [36 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 397 | 393 | 790

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or date last known alive. Survival data reflects the database as of December 23, 2013.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; every 6 months if patient is 2 - 5 years from study entry; then annually if patient is 5 - 10 years from study entry
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Number analyzed (Participants) | 397 | 393
months | 57.6 [49.1 to 72.8] | 44.0 [34.4 to 49.1]
Statistical Analysis 1: Comparison: Androgen-Deprivation Therapy and Docetaxel vs Androgen-Deprivation Therapy Alone; The study was designed to detect a 33.3% improvement in median survival time across treatments with one-sided type I error of 0.025 and 80% power; Test type: Superiority or Other; p = 0.0003, Log Rank

2. Secondary Outcome: Time to Clinical Progression
Description: Time to clinical progression is defined as the time from randomization to clinical progression. Clinical progression is defined as increasing symptomatic bone metastases, progression per Response Evaluation Criteria In Solid Tumors (RECIST) criteria or clinical deterioration due to cancer per investigator's opinion. Patients without documented clinical progression were censored at the date of last disease assessment. Secondary endpoint data reflect the database as of December 23, 2014.
Time Frame: as for outcome 1
Population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Number analyzed (Participants) | 397 | 393
months | 33.0 [27.3 to 41.2] | 19.8 [17.9 to 22.8]
Statistical Analysis 1: Comparison: Androgen-Deprivation Therapy and Docetaxel vs Androgen-Deprivation Therapy Alone; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Secondary Outcome: Time to Castration Resistant Prostate Cancer (Hormone Refractory Disease)
Description: Time to castration resistant prostate cancer is defined as the time from randomization to PSA progression or clinical progression, whichever occurred first. Patients without documented progression were censored at the date of last disease assessment. Secondary endpoint data reflect the database as of December 23, 2014.
Time Frame: as for outcome 1
Population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Number analyzed (Participants) | 397 | 393
months | 20.2 [17.2 to 23.6] | 11.7 [10.8 to 14.7]
Statistical Analysis 1: Comparison: Androgen-Deprivation Therapy and Docetaxel vs Androgen-Deprivation Therapy Alone; Test type: Superiority or Other; p < 0.0001, Log Rank

4. Secondary Outcome: Proportion of Patients With PSA Complete Response (CR) at 6 Months
Description: PSA CR is defined as a PSA level less than 0.2 ng/ml measured for 2 consecutive measurements at least 4 weeks apart. Patients who met the criterion of PSA CR and had PSA level less than 0.2 ng/ml before and after the 6-month time point are considered as having a PSA CR at 6 months.
Time Frame: Assessed at 6 months
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Number analyzed (Participants) | 397 | 393
proportion of participants | 0.320 [0.274 to 0.369] | 0.196 [0.158 to 0.239]
Statistical Analysis 1: Comparison: Androgen-Deprivation Therapy and Docetaxel vs Androgen-Deprivation Therapy Alone; Test type: Superiority or Other; p < 0.0001, Fisher Exact

5. Secondary Outcome: Proportion of Patients With PSA Complete Response (CR) at 12 Months
Description: PSA CR is defined as a PSA level less than 0.2 ng/ml measured for 2 consecutive measurements at least 4 weeks apart. Patients who met the criterion of PSA CR and had PSA level less than 0.2 ng/ml before and after the 12-month time point are considered as having a PSA CR at 12 months.
Time Frame: Assessed at 12 months
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Number analyzed (Participants) | 397 | 393
proportion of participants | 0.277 [0.234 to 0.324] | 0.168 [0.132 to 0.209]
Statistical Analysis 1: Comparison: Androgen-Deprivation Therapy and Docetaxel vs Androgen-Deprivation Therapy Alone; Test type: Superiority or Other; p < 0.0001, Fisher Exact

6. Secondary Outcome: QOL Change From Baseline to 3 Months
Description: The primary QOL change was evaluated by the Functional Assessment of Cancer Therapy - Prostate (FACT-P) instrument. FACT-P is a self-report measure of both general and disease-specific QOL. Higher scores represent better QOL. The FACT-P (version 4) contains 39 likert items distributed over 5 subscales: physical (7 items), social/family (7 items), emotional (6 items), and functional (7 items) well-being, and the additional concerns related to prostate cancer scale (12 items). The FACT-P total score is calculated by summing all these 5 subscales and ranges from 0 to 156.
Time Frame: Assessed at baseline and 3 months
Population: Patients with both baseline and 3-month QOL assessments are included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Androgen-Deprivation Therapy and Docetaxel | Androgen-Deprivation Therapy Alone
Number analyzed (Participants) | 334 | 299
units on a scale | -2.7 (0.9) | -1.1 (1.0)
Statistical Analysis 1: Comparison: Androgen-Deprivation Therapy and Docetaxel; Test type: Superiority or Other; p = 0.0009, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Androgen-Deprivation Therapy Alone; Test type: Superiority or Other; p = 0.40, Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Description: Submission of late adverse events is required at follow-up visits up to 10 years.
Groups:
- Arm A: Patients receive androgen-deprivation therapy (including luteinizing hormone-releasing hormone [LHRH] agonist therapy, LHRH antagonist therapy, or surgical castration). Patients also receive docetaxel IV over 1 hour on day 1. Treatment with docetaxel repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm B: Patients receive androgen-deprivation therapy (including luteinizing hormone-releasing hormone [LHRH] agonist therapy, LHRH antagonist therapy, or surgical castration).
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 116/390 | 12/392
Other Adverse Events (participants affected / at risk) | 38/390 | 1/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=390) | Arm B (N=392)
Allergic reaction (Immune system disorders) | 8 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 1
Leukocytes decreased (Investigations) | 18 | 0
Lymphopenia (Investigations) | 9 | 0
Neutrophils decreased (Investigations) | 47 | 0
Platelets decreased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 16 | 1
Weight gain (Investigations) | 2 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0
Skin-other (Skin and subcutaneous tissue disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 1
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 24 | 0
Infection w/ gr3-4 neut, heart (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, skin (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 2 | 0
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, rectum (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, blood (Infections and infestations) | 1 | 0
Infection-other (Infections and infestations) | 1 | 0
Edema limb (General disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Neuropathy-motor (Nervous system disorders) | 2 | 0
Neuropathy-sensory (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Cardiac/heart, pain (Cardiac disorders) | 1 | 0
Head/headache (Nervous system disorders) | 0 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erectile impotence (Reproductive system and breast disorders) | 1 | 2
Gynecomastia (Reproductive system and breast disorders) | 1 | 1
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=390) | Arm B (N=392)
Fatigue (General disorders) | 35 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less